CLINICAL TRIAL: NCT04478994
Title: A Randomized, Double-Blind, Placebo-Controlled, Repeat-Dose, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics, and Explore Efficacy of TEPEZZA in Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: A Study With TEPEZZA in Patients With Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-TEP-001
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — teprotumumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEPEZZA 20mg/kg (Active Comparator): Approximately 15 participants will receive 8 infusions of TEPEZZA q3W for a total of 21 weeks. TEPEZZA 10mg/kg will be administered on Day 1 and TEPEZZA 20mg/kg will be administered q3W for the remaining 7 infusions.
  Interventions: Biological: TEPEZZA
- Placebo (Placebo Comparator): Approximately 10 participants will receive 8 infusions of placebo q3W for a total of 21 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TEPEZZA — TEPEZZA is a fully human anti-IGF-1R mAb. TEPEZZA will be provided in single-dose 20 mL glass vials as a freeze-dried powder. Each vial of TEPEZZA must be reconstituted with 10 mL of water for injection. Reconstituted TEPEZZA solution must be further diluted in 0.9% (w/v) sodium chloride (NaCl) solution prior to administration. TEPEZZA will be administered in 100 mL or 250 mL infusion bags (100 mL infusion bags for doses up to 1800 mg and 250 mL infusion bags for doses > 1800 mg).
  Other Names: teprotumumab-trbw; HZN-001
  Arms: TEPEZZA 20mg/kg
Other: Placebo — Placebo will consist of normal saline (0.9% NaCl) solution and will be administered in 100 mL or 250 mL infusion bags, as would be appropriate, per weight-based dosing volumes (100 mL infusion bags for doses up to 1800 mg and 250 mL infusion bags for doses > 1800 mg).
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The overall objective is to investigate the safety, tolerability and effect on insulin-like growth factor-1 (IGF-1), inflammatory and fibrotic biomarkers of TEPEZZA (teprotumumab-trbw, HZN-001), a fully human monoclonal antibody (mAb) inhibitor of the IGF-1 receptor (IGF-1R), administered once every 3 weeks (q3W) for 24 weeks in the treatment of participants with diffuse cutaneous systemic sclerosis (dcSSc).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, repeat-dose, multicenter study. Participants will be screened for the study within 4 weeks prior to the Baseline (Day 1) Visit. Approximately 25 participants who meet the study eligibility criteria will be randomized on Day 1 in a 3:2 ratio to receive 8 infusions of TEPEZZA or placebo q3W. During the 24-week double-blind Treatment Period, study drug will be infused on Day 1 (Baseline) and Weeks 3, 6, 9, 12, 15, 18 and 21 with a comprehensive visit at Week 24 (end of treatment). On each dosing day, scheduled assessments (except for Adverse Events [AE] and concomitant medication use monitoring, which will be monitored throughout the clinic visit) will be completed prior to study drug infusions.

At the end of the Treatment Period (Week 24), participants will enter a 24-week Follow-up Period, during which study drug will not be administered and a clinic visit will be scheduled for Weeks 28, 36 and 48. A phone call or email at Weeks 32 and 42 will occur to inquire how the participant is doing.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female between the ages of 18 and 80 years, inclusive, at Screening.
3. Meets the 2013 American College of Rheumatology/European League Against Rheumatism classification criteria for systemic sclerosis (SSc) with a total score of ≥9.
4. Classified as having skin involvement proximal to elbow, knee, face and neck.
5. At the time of enrollment, no more than 60 months must have elapsed since the onset of the first dcSSc manifestations, other than Raynaud's phenomenon.
6. Skin thickening from dcSSc in the forearm suitable for repeat biopsy.
7. Modified Rodman Skin Score (mRSS) units ≥10 and ≤45 at Screening.
8. Participant will be allowed to take CellCept® (mycophenolate mofetil) up to 3 g/day or Myfortic® (mycophenolic acid) up to 2.14 g/day and low-dose prednisone (≤10 mg/day or equivalent dosing of glucocorticoids). Participants taking CellCept or Myfortic have been doing so for ≥20 weeks and the dose must have been stable for ≥16 weeks prior to the Day 1 Visit. Prednisone must have been at a stable dose for ≥4 weeks prior to the Day 1 Visit.
9. Diabetic participants must have glycated hemoglobin (HbA1c) ≤8.0%, with no new diabetic medication (oral or insulin) or more than a 10% change in the dose of a currently prescribed diabetic medication within 60 days prior to Screening.
10. Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, nontherapy-induced amenorrhea for <12 months prior to Screening or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified timepoints (i.e., prior to each dose and throughout the participant's participation in the Follow-up Period); participants who are sexually active with a non vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least one full cycle prior to Baseline and continue for 180 days after the last dose of study drug. Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner.
11. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.

Exclusion Criteria:

1. Diagnosed with limited cutaneous SSc or sine scleroderma.
2. Diagnosed with other autoimmune connective tissue diseases, except for fibromyalgia, scleroderma associated myopathy and Sjogren's syndrome.
3. Scleroderma renal crisis diagnosed within 6 months of the Screening Visit, characterized by abrupt onset of hypertension and acute kidney injury.
4. Forced vital capacity (FVC) <50% predicted, diffusing capacity of the lungs for carbon monoxide (DLCO) <40% predicted or pulmonary arterial hypertension (PAH) by right heart catheterization requiring treatment with more than one oral PAH approved therapy or parenteral therapy (intermittent use of phosphodiesterase-5 inhibitors are allowed for erectile dysfunction and/or Raynaud's phenomenon/digital ulcers).
5. Corticosteroid use for conditions other than dcSSc within 4 weeks prior to Screening (topical steroids for dermatological conditions and inhaled steroids are allowed).
6. Previous treatment with rituximab (Rituxan® or MabThera®) within 12 months prior to the first infusion.
7. Use of a non-steroidal immunosuppressive agent, cytotoxic or anti-fibrotic drug within 4 weeks of Screening, including cyclophosphamide, azathioprine (Imuran®), methotrexate or other immunosuppressive or cytotoxic medication. Exceptions are mycophenolate mofetil (CellCept) and mycophenolic acid (Myfortic), which are permitted according to inclusion criterion 8, and anti-malarials (e.g., hydroxychloroquine [Plaquenil®]).
8. Use of biologics or small molecules approved for rheumatoid arthritis, psoriatic arthritis and other rheumatic diseases within 4 weeks prior to Screening.
9. Use of an investigational agent for any condition within 90 days or 5 half-lives, whichever is longer, prior to Screening or anticipated use during the course of the trial.
10. Malignant condition in the past 5 years (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
11. Pregnant or lactating women.
12. Current drug or alcohol abuse or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the participant.
13. Biopsy-proven or clinically suspected inflammatory bowel disease (e.g., diarrhea with or without blood or rectal bleeding associated with abdominal pain or cramping/colic, urgency, tenesmus or incontinence for more than 4 weeks without a confirmed alternative diagnosis OR endoscopic or radiologic evidence of enteritis/colitis without a confirmed alternative diagnosis).
14. Known hypersensitivity to any of the components of TEPEZZA or prior hypersensitivity reactions to mAbs.
15. Previous enrollment in this study or participation in a prior teprotumumab-trbw clinical trial.
16. Human immunodeficiency virus, untreated or positive viral load for hepatitis C or hepatitis B infections.
17. Previous organ transplant (including allogeneic and autologous marrow transplant).
18. Alanine aminotransferase or aspartate aminotransferase >2.5 times the upper limit of normal or estimated glomerular filtration rate of <30 mL/min/1.73m^2 at Screening.
19. Platelets <100×10^3/µL.
20. Hemoglobin <8 g/dL.
21. Any other condition that, in the opinion of the Investigator, would preclude inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - UCLA Division of Rheumatology, Los Angeles, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - Yale North Haven Medical Center, New Haven, Connecticut
  - The Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - UT Physicians Center for AutoImmunity, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Groups:
- TEPEZZA 20 mg/kg: Participants receive 8 infusions of TEPEZZA every 3 weeks (q3W) for a total of 21 weeks: TEPEZZA 10 mg/kg administered on Day 1 and TEPEZZA 20 mg/kg administered q3W for the remaining 7 infusions.
- Placebo: Participants receive 8 infusions of placebo q3W for a total of 21 weeks.
Period: Overall Study
Arm/Group | TEPEZZA 20 mg/kg | Placebo
Started | 1 | 2
Completed | 0 | 1
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEPEZZA 20 mg/kg | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Treatment Emergent Adverse Event (TEAE) Through Week 24
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. TEAEs are those that occurred after the first dose of trial drug.
Time Frame: From first dose of trial drug up to Week 24
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | TEPEZZA 20 mg/kg | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: From enrollment (all-cause mortality) or first dose of trial drug on Day 1 (adverse events) until 3 weeks (21 days) after last dose of trial drug, up to Week 48.
Arm/Group | TEPEZZA 20 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEPEZZA 20 mg/kg (N=1) | Placebo (N=2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEPEZZA 20 mg/kg (N=1) | Placebo (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Weight decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04478994/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04478994/SAP_001.pdf